CLINICAL TRIAL: NCT03438942
Title: The Study of the Influence of Intestinal and Cellular Iron and Foliate Transporters on Bioavailability of These Micronutrients in the Organism
Brief Title: Influence of Iron and Foliate Transporters on Bioavailability of These Micronutrients in the Organism
Acronym: WiMKo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Life Sciences (Other)
Responsible Party: Principal Investigator, Joanna Suliburska, assistant professor, Poznan University of Life Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 917/16
Record Dates: First submitted 2018-02-13; First posted 2018-02-20 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Nutrition Disorders
Keywords: iron; folate; childbearing age; bioavailability
MeSH Terms: conditions — Nutrition Disorders | interventions — Folic Acid; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Folic acid and iron supplementation (Experimental): Individuals with low level of blood folic acid and iron- will receive folic acid and iron supplementation daily, for 3 months
  Interventions: Dietary Supplement: Folic acid and iron supplementation
- Control group (Active Comparator): Individuals with proper level of blood folic acid and iron- will not receive folic acid and iron supplementation daily, for 3 months
  Interventions: Dietary Supplement: Control group

INTERVENTIONS:
Dietary Supplement: Folic acid and iron supplementation — Individuals with low level of blood folic acid and iron- will receive folic acid and iron supplementation daily, for 3 months
  Arms: Folic acid and iron supplementation
Dietary Supplement: Control group — Individuals with proper level of blood folic acid and iron- will not receive folic acid and iron supplementation daily, for 3 months
  Arms: Control group

SUMMARY:
The aim of the study is to determine the factors affecting the bioavailability of iron and folic acid during the simultaneous use of iron supplements and folic acid supplements in non-pregnant women of childbearing age.

DETAILED DESCRIPTION:
Scientists in the field of nutrition and gynecology and obstetrics have been paying attention to the need of use iron and folate supplements in women of childbearing age. Increased intake of micronutrients in the diet or the use of supplementation does not always bring the expected results, what depends on factors that affect the bioavailability of minerals and vitamins. On the one hand these factors are related to the properties of food intake, e.g. to the presence of other nutrients that can increase or decrease the absorption of folates and iron (eg vitamin C, phytates), and on the other hand the functioning of the body itself, which to a certain extent is determined by genetic factors (e.g., genetically determined reduced activity of methylenetetrahydrofolate reductase [MTHFR], which reduces the bioavailability of folic acid).

The study aims:

* assessment of the effect of simultaneous supplementation with iron and folate on:

  * parameters of the iron metabolism
  * parameters of the folate metabolism
* the estimation of gene polymorphisms encoding proteins transporting iron and folate
* obtaining information whether the polymorphism of genes encoding proteins transporting iron and folate is related to the effectiveness of the iron and folic acid supplementation used in non-pregnant women of childbearing age.

In 200 non-pregnant women of childbearing age a blood level of iron and folic acid will be determined. Subjects with low level of blood iron and folic acid will be supplemented with oral iron and folic acid for 3 months. Subjects with proper level of blood iron and folic acid will be a control group. At baseline and at completion of the study (after 3 months) fasting blood will be collected and abovementioned parameters will be estimated.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 35 years
* stable body weight (< 3 kg self-reported change during the previous three months)
* written informed consent to participate in the study,
* regular menstrual period;
* regular diet

Exclusion Criteria:

* history of use of any dietary supplements within the one month prior to the study containing iron or folic acid
* clinically relevant acute or chronic inflammatory disease in the respiratory, gastrointestinal or genitourinary system or in the mouth, throat, paranasal sinuses and / or connective tissue disease, arthritis;
* simultaneous participation in a study that affects body weight or use of diet / medication / nutritional behaviors affecting body weight;
* a history of infection in the month prior to the study
* nicotine, drug or alcohol abuse
* vegetarian diet;
* pregnancy or lactation
* other condition that, in the opinion of the investigators, would make participation not in the best interest of the patient or could prevent, limit, or confound the study results

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female gender based on self-representation
Enrollment: 200 (Actual)
Dates: Start 2018-09-30 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
folic acid concentrations at baseline | At the baseline
  blood folic acid concentrations at baseline
folic acid concentrations after 3 months of treatment | after 3 months of treatment
  blood folic acid concentrations after 3 months of treatment
iron concentrations at baseline | At the baseline
  blood iron concentrations at baseline
iron concentrations after 3 months of treatment | after 3 months of treatment
  blood ron concentrations after 3 months of treatment

SECONDARY OUTCOMES:
blood pressure | At the baseline
  blood pressure
body mass | At the baseline
  body mass
body height | At the baseline
  body height
Body % fat | At the baseline
  Fat tissue % estimated with air displacement plethysmography
Body % muscle | At the baseline
  Muscle tissue % estimated with BodPod (air displacement plethysmography)
ferritin at the baseline | At the baseline
  serum ferritin concentration at the baseline
ferritin after 3 months of treatment | after 3 months of treatment
  serum ferritin concentration after 3 months of treatment
hepcidin at the baseline | At the baseline
  serum hepcidin concentration at the baseline
hepcidin after 3 months of treatment | after 3 months of treatment
  serum hepcidin concentration after 3 months of treatment
homocysteine at the baseline | At the baseline
  serum homocysteine concentration at the baseline
homocysteine after 3 months of treatment | after 3 months of treatment
  serum homocysteine concentration after 3 months of treatment
total iron-binding capacity (TIBC) at the baseline | At the baseline
  Blood total iron-binding capacity at the baseline
TIBC after 3 months of treatment | after 3 months of treatment
  Blood total iron-binding capacity after 3 months of treatment
divalent metal transporter 1 (DMT1) gene polymorphisms | At the baseline
  polymorphisms of gene encoding divalent metal transporter 1
transferrin receptor 2 (TfR2) gene polymorphisms | At the baseline
  polymorphisms of gene encoding transferrin receptor 2
proton-coupled folate transporter (PCFT) gene polymorphisms | At the baseline
  polymorphisms of gene encoding proton-coupled folate transporter
reduced folate carrier (RFC) gene polymorphisms | At the baseline
  polymorphisms of gene encoding reduced folate carrier

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Suliburska, Ass Prof, Principal Investigator — Institute of Human Nutrition and Dietetics, Poznań University of Life Sciences
Locations (1):
- Poznan University of Life Sciences, Poznan, Poland